CLINICAL TRIAL: NCT02497729
Title: Checklists and Upright Positioning in Endotracheal Intubation of Critically Ill Patients (Check-UP) Trial
Acronym: Check-UP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Todd Rice, Associate Professor of Medicine, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 150897
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Respiratory Failure
Keywords: Endotracheal Intubation; Checklist; Positioning
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Checklist; Patient Positioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sniffing Position, No Checklist (No Intervention): Patient in the sniffing position without the use of a written checklist
- Sniffing Position, Checklist (Active Comparator): Patient in the sniffing position with the use of a written checklist
  Interventions: Procedure: Written Checklist
- Head of Bed Up, No Checklist (Active Comparator): Patient with the head of bed up and without the use of a checklist
  Interventions: Procedure: Head of Bed Up
- Head of Bed Up, Checklist (Active Comparator): Patient with the head of bed up and with the use of a checklist
  Interventions: Procedure: Written Checklist; Procedure: Head of Bed Up

INTERVENTIONS:
Procedure: Written Checklist — Use of a written checklist pre and peri-intubation
  Other Names: Checklist
  Arms: Head of Bed Up, Checklist; Sniffing Position, Checklist
Procedure: Head of Bed Up — Raising the patient's head of bed to 25 degrees
  Other Names: Patient Positioning; Sniff Position
  Arms: Head of Bed Up, Checklist; Head of Bed Up, No Checklist

SUMMARY:
The use of a written, pre-procedure checklist and positioning the patient with the head of the bed elevated have been proposed as interventions capable of preventing complications during non-elective intubation and are used intermittently in routine care -- however neither have been examined in a prospective trial.

DETAILED DESCRIPTION:
Endotracheal intubation is common in the care of critically ill patients. Procedural complications including hypoxia and hypotension are frequent in urgent and emergent intubation and associated with an increased risk of death. The use of a written, pre-procedure checklist and positioning the patient with the head of the bed elevated have been proposed as interventions capable of preventing complications during non-elective intubation and are used intermittently in routine care -- however neither have been examined in a prospective trial. The investigators propose a randomized trial comparing use of a written checklist versus no written checklist and ramped versus sniffing position for endotracheal intubation of critically ill adults.

ELIGIBILITY:
Inclusion Criteria:

Airway management events will be included in which:

1. Patient is admitted to the Medical Intensive Care Unit (MICU)
2. Planned procedure is endotracheal intubation
3. Planned operator is a Pulmonary and Critical Care Medicine (PCCM) fellow
4. Administration of sedation and/or neuromuscular blockade is planned
5. Age ≥ 18 years old

Exclusion Criteria:

Airway management events will be excluded in which:

1. Operator feels specific patient positioning during intubation is required
2. Urgency of intubation precludes safe performance of study procedures
3. Operator feels an alternative pre-procedure checklist or no checklist is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Lowest Arterial Oxygen Saturation (Both positioning and Checklist interventions) | Time of Induction through 2 minutes after successful intubation
  Lowest non-invasively measured arterial oxygen saturation between the time of induction or neuromuscular blockade and two minutes after completion of the airway management procedure
Lowest Systolic Blood Pressure (Checklist intervention only) | Time of Induction through 2 minutes after successful intubation
  Lowest non-invasively or invasively measured systolic blood pressure between medication administration and 2 minutes following successful placement of an endotracheal tube (in checklist comparison only)

SECONDARY OUTCOMES:
Incidence of Desaturation | Time of Induction through 2 minutes after successful intubation
  Decrease in oxygen saturation of greater than 3% from induction to lowest oxygen saturation
Incidence of Hypoxemia | Time of Induction through 2 minutes after successful intubation
  Defined by lowest oxygen saturation less than 90% and severe hypoxemia as defined by lowest oxygen saturation less than 80%
Change in Saturation | Time of Induction through 2 minutes after successful intubation
  Change in oxygen saturation from baseline to lowest oxygen saturation
Grade of First Glottic View | Time of Induction through 2 minutes after successful intubation
  Cormack-Lehane grade of view on first intubation attempt
First Pass Success | Time of Induction through 2 minutes after successful intubation
  Placement of an endotracheal tube in the trachea after the first insertion of the laryngoscope into the oral cavity without the use of any other devices
Number of Intubation Attempts | Time of Induction through 2 minutes after successful intubation
  Number of attempts required for successful tube placement
Time to Intubation | Time of Induction through 2 minutes after successful intubation
  Time (in minutes) from pushing of induction meds to successful placement of endotracheal tube
Need for Assistance | Time of Induction through 2 minutes after successful intubation
  Incidence of need for additional intubating equipment, second operator
Non-hypoxic complications | Time of Induction through 2 minutes after successful intubation
  Incidence of non-oxygenation complications - composite of all other recorded complications
Malposition of Endotracheal Tube | Time of Induction through 2 minutes after successful intubation
  Incidence of post-intubation tube malposition on Chest X-Ray (CXR)
Repositioning Patient | Time of Induction through 2 minutes after successful intubation
  Incidence of repositioning patient after procedure initiation
In-Hospital Mortality | From enrollment through the earlier of hospital discharge or 365 days
  Death before hospital discharge
Ventilator-free Days | From enrollment through study day 28
  Days alive and free from mechanical ventilation
ICU-Free Days | From enrollment through study day 28
  Days alive and out of the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Todd W Rice, MD, MSc, Study Director — Vanderbilt University Medical Center
Locations (5):
- United States (5):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Vanderbilt University, Nashville, Tennessee
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Janz DR, Semler MW, Joffe AM, Casey JD, Lentz RJ, deBoisblanc BP, Khan YA, Santanilla JI, Bentov I, Rice TW; Check-UP Investigators*; Pragmatic Critical Care Research Group. A Multicenter Randomized Trial of a Checklist for Endotracheal Intubation of Critically Ill Adults. Chest. 2018 Apr;153(4):816-824. doi: 10.1016/j.chest.2017.08.1163. Epub 2017 Sep 14. PMID 28917549
- [Derived] Semler MW, Janz DR, Russell DW, Casey JD, Lentz RJ, Zouk AN, deBoisblanc BP, Santanilla JI, Khan YA, Joffe AM, Stigler WS, Rice TW; Check-UP Investigators( *); Pragmatic Critical Care Research Group. A Multicenter, Randomized Trial of Ramped Position vs Sniffing Position During Endotracheal Intubation of Critically Ill Adults. Chest. 2017 Oct;152(4):712-722. doi: 10.1016/j.chest.2017.03.061. Epub 2017 May 6. PMID 28487139